CLINICAL TRIAL: NCT02106520
Title: Efficacy of a Bevacizumab Nasal Spray as a Treatment for Epistaxis in Hereditary Hemorrhagic Telangiectasia (HHT)
Acronym: ALEGORI
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: DSMB's decision following the first step analysis
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2013.827
Record Dates: First submitted 2014-04-01; First posted 2014-04-08 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-11

CONDITIONS: Hereditary Hemorrhagic Telangiectasia; Epistaxis
Keywords: Epistaxis; Bevacizumab
MeSH Terms: conditions — Telangiectasia, Hereditary Hemorrhagic; Epistaxis | interventions — Bevacizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Bevacizumab 25mg (Experimental): Three administrations of 25 mg of Bevacizumab spaced of 14 days
  Interventions: Drug: Bevacizumab
- Bevacizumab 50mg (Experimental): Three administrations of 50 mg of Bevacizumab spaced of 14 days
  Interventions: Drug: Bevacizumab
- Bevacizumab 75mg (Experimental): Three administrations of 75 mg of Bevacizumab spaced of 14 days
  Interventions: Drug: Bevacizumab
- Placebo (Placebo Comparator): Three administrations of placebo spaced of 14 days
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Bevacizumab
  Other Names: Three administrations of Bevacizumab spaced of 14 days
  Arms: Bevacizumab 25mg; Bevacizumab 50mg; Bevacizumab 75mg
Drug: placebo
  Other Names: Three administrations of placebo spaced of 14 days
  Arms: Placebo

SUMMARY:
Hereditary Hemorrhagic Telangiectasia (HHT) is a rare (~ 1/6000) but ubiquitous genetic disease. It is associated with abnormal angiogenesis and autosomal dominant inheritance, leading to telangiectasias and arteriovenous fistulae. More than 95% of patients are concerned by epistaxis (nosebleeds). These events are spontaneous, repeated, irregular, both diurnal and nocturnal, a source of anemia, disabling and very socially embarrassing.

Anti-angiogenic treatments, including bevacizumab, are a new therapeutic option in HHT.

The aim of this study is to evaluate 3 months after the end of the treatment the efficacy on the duration of the nosebleeds with 3 different doses (25, 50 and 75 mg) of bevacizumab administered as a nasal spray in a repeated manner (3 administrations) in patients with Hereditary Hemorrhagic Telangiectasia complicated by nosebleeds.

This randomized, double-blind, placebo-controlled, seamless phase II/III study is to be carried out on 4 groups of 20 patients for first step and 2 groups of 20 to 40 patients for second step

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Patients who have given their free informed and signed consent.
* Patients affiliated to a social security scheme or similar.
* Patients monitored for clinically confirmed HHT (presence of at least 3 Curaçao criteria) and/or confirmed by molecular biology.
* Patients who have not undergone nasal surgery in the 3 months prior to inclusion.
* Patient with nosebleeds of a monthly duration of more than 20 minutes and justified by follow-up grids completed for at least the 3 months prior to the time of inclusion.

Exclusion Criteria:

* Women who are pregnant or likely to become so in the course of the study.
* Patients not affiliated to a social security scheme.
* Patients who are protected adults under the terms of the law (French Public Health Code).
* Refusal to consent.
* Patients for whom the diagnosis of HHT has not been confirmed clinically and/or by molecular biology.
* Patients with an on-going infectious condition.
* Participation in another clinical trial within the 28 days prior to inclusion.
* Known hypersensitivity to the active ingredient or one of the excipients.
* Known hypersensitivity to products of Chinese hamster ovary cells (CHO) or other human or humanized recombinant antibodies.
* Patients who have incompletely filled in the nosebleed grids in the 3 months preceding the treatment.
* Patients who do not present with nosebleeds with a monthly average duration over the 3 months preceding the treatment of more than 20 minutes ((duration M1 + duration M2 + duration M3) / 3). Remark: only the 3 months strictly preceding the treatment will be taken into account, even if the grids have been completed over a longer period.
* Patients who have received Avastin® intravenously in the 6 months prior to inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2014-04; Primary Completion 2015-06 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
mean duration of epistaxis | 3 months after treatment
  To evaluate 3 months after the end of the treatment the efficacy on the duration of the nosebleeds with 3 different doses (25, 50 and 75 mg) of bevacizumab administered as a nasal spray in a repeated manner (3 administrations).

SECONDARY OUTCOMES:
adverse events | before and 6 months after treatment
  Adverse events observed along a repeated administration of bevacizumab (nasal spray administration) : evaluation by epistaxis monitoring along the study and by a clinical exam before each treatment and 6 months after the end of the treatment.
mean monthly epistaxis duration | 6 months after the end of the treatment
  To evaluate the efficacy at 6 months after the end of the treatment on the duration of the nosebleeds for the dose retained versus placebo
frequency and duration of epistaxis | 3 months and 6 months after the end of the treatment
  Evolution of the frequency and the mean monthly duration of epistaxis at 3 and 6 months for the dose retained
Quality of life | 3 months and 6 months aftert the end of the treatment
  Evolution of the quality of life score (SF-36) between the inclusion, 3 months and 6 months after the end of the treatment
Number of red blood cells transfusion | 3 months and 6 months after the end of the treatment
  Evolution of the number of red blood cells transfusion between the inclusion and 3 and 6 months after the end of the treatment.
Change in hemoglobinemia and serum ferritin | 1 month, 3 months and 6 months
  Evolution of hemoglobinemia and serum ferritin at inclusion,3 and 6 months after the end of the treatment for the retained dose
Kinetics of monthly epistaxis duration | 6 months
  To describe the nosebleed kinetics for the dose retained and the placebo throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Sophie DUPUIS-GIROD, MD, Principal Investigator — Service de génétique, Hôpital Louis Pradel, Hospices Civils de Lyon
Locations (1):
- Hôpital Louis Pradel, Bron, France

REFERENCES:
- [Derived] Dupuis-Girod S, Ambrun A, Decullier E, Fargeton AE, Roux A, Breant V, Colombet B, Riviere S, Cartier C, Lacombe P, Chinet T, Blivet S, Blondel JH, Gilbert-Dussardier B, Dufour X, Michel J, Harle JR, Dessi P, Faure F. Effect of Bevacizumab Nasal Spray on Epistaxis Duration in Hereditary Hemorrhagic Telangectasia: A Randomized Clinical Trial. JAMA. 2016 Sep 6;316(9):934-42. doi: 10.1001/jama.2016.11387. PMID 27599328